CLINICAL TRIAL: NCT01019655
Title: Low Molecular Weight Heparin for Pregnant Women With Thrombophilia: a Prospective, Randomized, Open Trial
Brief Title: Heparin for Pregnant Women With Thrombophilia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Clemens Tempfer, MD, University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: tempfer2.0
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Pregnancy and Thrombophilia
Keywords: thrombophilia; pregnancy; heparin
MeSH Terms: conditions — Thrombophilia | interventions — Nadroparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nadroparin calcium (Experimental): nadroparin calcium (fraxiparin®) 0.3 mL daily during pregnancy and six weeks post partum
  Interventions: Drug: Nadroparin calcium
- Control (No Intervention): No intervention other than usual care at the study site

INTERVENTIONS:
Drug: Nadroparin calcium — nadroparin calcium (fraxiparin®) 0.3 mL daily during pregnancy and six weeks post partum
  Other Names: Fraxiparin; code number EU:1-21067
  Arms: Nadroparin calcium

SUMMARY:
The purpose of this study is to investigate whether heparin is an effective treatment in pregnant women at risk for thrombosis and other pregnancy-associated complications.

DETAILED DESCRIPTION:
Women with thrombophilia, i.e. carriage of a factor V leiden mutation, a factor II prothrombin G20210A mutation or a reduced amount of antithrombin III, protein C or protein S, are at elevated risk for thrombosis and related sequelae. Specifically, pregnant women with thrombophilia are at risk for pregnancy-associated thrombosis, pregnancy-associated thromboembolism as well as early miscarriage (until 20 weeks gestation) late miscarriage (after 20 weeks gestation), preeclampsia, and intrauterine growth retardation <10th percentile. Uncontrolled retrospective and prospective studies indicate that a therapy with unfractionated heparin or low molecular weight heparin in pregnancy significantly reduces these pregnancy complications and improves maternal and fetal outcome. The use of low molecular weight heparin in pregnancy is safe with complication rates between 1% and 3%, mainly thrombocytopenia and bleeding complications. Randomized trials to adequately assess the safety and efficacy of heparin in pregnant women with thrombophilia are not available to date. Thus, we intend to randomize pregnant women with thrombophilia during weeks of gestation 11 to 14 into a therapy with nadroparin calcium (fraxiparin®) 0.3 mL daily during pregnancy and six weeks post partum and usual care. The primary end point of this study is a composite endpoint of pregnancy-associated thrombosis, pregnancy-associated thromboembolism, early miscarriage (until 20 weeks gestation) late miscarriage (after 20 weeks gestation), preeclampsia, and intrauterine growth retardation <10th percentile. We hypothesize that a prophylactic therapy with nadroparin calcium will significantly reduce pregnancy complications in pregnant women with thrombophilia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a singleton pregnancy
* Age >18 years
* Ability to understand informed consent form

Exclusion Criteria:

* Allergy/hypersensitivity for nadroparin calcium
* Heparin-associated thrombocytopenia
* Organ lesions at risk for bleeding such as acute stomach/bowel ulcers, cerebral hemorrhage, cerebral aneurysm
* uncontrolled hypertension
* Liver and/or renal dysfunction
* Known hematologic disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
composite endpoint: pregnancy-associated thrombosis/thromboembolism, miscarriage, preeclampsia, intrauterine growth retardation | 10.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Clemens B Tempfer, MD, Principal Investigator — University of Vienna
Locations (1):
- Department of Obstetrics and Gynecology, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Middleton P, Shepherd E, Gomersall JC. Venous thromboembolism prophylaxis for women at risk during pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2021 Mar 29;3(3):CD001689. doi: 10.1002/14651858.CD001689.pub4. PMID 33779986
- [Derived] Bennett SA, Bagot CN, Arya R. Pregnancy loss and thrombophilia: the elusive link. Br J Haematol. 2012 Jun;157(5):529-42. doi: 10.1111/j.1365-2141.2012.09112.x. Epub 2012 Mar 26. PMID 22449204